CLINICAL TRIAL: NCT03996434
Title: Coasting Versus Gonadotrophin-Releasing Hormone Antagonist Administration in Patients at High Risk of Ovarian Hyperstimulation Syndrome and Its Impact on the Embryos Quality and the Outcome of ICSI
Brief Title: Coasting Versus Antagonist Protocol in Patients at High Risk of OHSS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ClinAmygate (Other)
Collaborators: Cairo University (Other); Al-Azhar University (Other); Beni-Suef University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Clin-I-0201907
Record Dates: First submitted 2019-06-21; First posted 2019-06-24 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Ovarian Hyperstimulation Syndrome
MeSH Terms: conditions — Ovarian Hyperstimulation Syndrome | interventions — Gonadotropins; cetrorelix

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coasting group (Experimental): Including 150 patients who will undergo withholding gonadotropin administration for at least 24 hours before triggering ovulation with hCG. GnRH agonist will be continued daily till the day of triggering. E2 will be measured daily until the concentration falls to ≤ 3000 pg/ml, then 5000 IU of hCG will be given.
  Interventions: Drug: Gonadotropin
- Antagonist group (Active Comparator): Including 150 patients who will receive GnRH antagonist (subcutaneous injection Cetrorelix acetate 0.25 mg (Cetrotide, Serono, UK)) daily until the day of hCG administration.
  GnRH agonist will be discontinued at the start of antagonist administration.
  E2 will be measured daily until the concentration falls to ≤ 3000 pg/ml and TVS revealed that follicles diameter is ≥ 18 mm, then 5000 IU of hCG will be given.
  Interventions: Drug: Antagonist

INTERVENTIONS:
Drug: Gonadotropin — withholding gonadotropin administration for at least 24 hours
  Arms: Coasting group
Drug: Antagonist — Cetrorelix acetate 0.25 mg
  Other Names: Cetrorelix acetate
  Arms: Antagonist group

SUMMARY:
The aim of this work is to study the value of GnRH antagonist subcutaneous administration as an alternative to coasting in prevention of severe OHSS and its impact on embryos quality & the outcome of ICSI.

DETAILED DESCRIPTION:
Infertility affects up to one in seven couples all over the world. In vitro fertilization-embryo transfer (IVF-ET) and intracytoplasmic sperm injection (ICSI) are commonly used in the management of infertility attributable to tubal factor, significant endometriosis, male factor and also persistent unexplained infertility. Recruitment and development of multiple follicles in response to gonadotrophin stimulation are necessary for successful assisted reproduction. In young ovulating women undergoing IVF treatment, the standard stimulation protocol can result in either poor response or ovarian hyperstimulation syndrome (OHSS).

OHSS is a serious and potentially life-threatening iatrogenic complication of controlled ovarian hyperstimulation (COH) which may cause serious impact on patient's health. OHSS is the most feared complication of IVF-related ovarian stimulation, which in its severe form leads to hospitalization and in the worst case scenario fatal complications. As many as 33% of IVF cycles have been reported to be associated with mild forms of OHSS. The incidence of moderate OHSS is estimated to be between 3% and 6%, while the severe form may occur in 0.1-3% of all cycles. Among high risk women the incidence approaches 20%.

Development of multiple follicles forms the basis of OHSS. Exogenous human chorionic gonadotrophin (hCG) administration for the final maturation of oocytes or endogenous production of hCG after pregnancy is the second factor needed for the development of severe OHSS. Severe OHSS is characterized by massive ovarian enlargement, pleural effusion, ascites, oliguria, hemoconcentration, and thromboembolic phenomena. Coasting is described as a withholding therapy while continuing with releasing hormone agonist/antagonist administration, until safe levels of estradiol (E2) are attained. GnRH antagonists causes an immediate suppression of E2 levels and therefore could prevent OHSS in GnRH antagonist cycles. A comparison between coasting and GnRH antagonist administration in women at high risk of OHSS during ovarian stimulation for IVF with GnRH agonist long protocol, in the hope of preventing the drawbacks of prolonged coasting.

ELIGIBILITY:
Inclusion Criteria:

* infertile women
* age 20-40
* at high risk for OHSS

Exclusion Criteria:

* refuse to participate

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 300 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-11-10 (Actual); Study Completion 2019-11-20 (Actual)

PRIMARY OUTCOMES:
Number of high quality embryos | Within 48 hours of fertilization
  Number of high quality embryos

CONTACTS AND LOCATIONS:
Overall Officials: Eman Elgendy, MD, Principal Investigator — International Islamic Centre for Population Studies and Research
Locations (2):
- Egypt (2):
  - Alazahr University, Cairo
  - Assisted Reproduction Unit International Islamic Centre for Population Studies and Research, Al-Azhar University, Cairo

IPD SHARING:
Plan to Share IPD: No
Local regulations

REFERENCES:
- [Result] Aboulghar MA, Mansour RT, Amin YM, Al-Inany HG, Aboulghar MM, Serour GI. A prospective randomized study comparing coasting with GnRH antagonist administration in patients at risk for severe OHSS. Reprod Biomed Online. 2007 Sep;15(3):271-9. doi: 10.1016/s1472-6483(10)60339-2. PMID 17854523